CLINICAL TRIAL: NCT00246506
Title: Optimal Infertility Therapy RCT: Women 40 and Older
Brief Title: Infertility Therapy for Women Age Thirty-eight and Older
Acronym: FORT-T
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R01HD044547 (NIH)
Record Dates: First submitted 2005-10-27; First posted 2005-10-31 (Estimated); Last update posted 2013-01-15 (Estimated); Status verified 2012-12

CONDITIONS: Infertility
Keywords: Infertility; Fertility; Reproduction; Advanced Maternal Age; Reproductive Medicine; Reproductive Techniques; Pregnancy
MeSH Terms: conditions — Infertility | interventions — Fertilization in Vitro; Reproductive Techniques, Assisted

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- I. (Active Comparator): Those randomized to have clomiphene/IUI treatments first will initiate therapy with two cycles of the fertility pill called clomiphene combined with (IUI) intrauterine insemination. If not pregnant after 2 IUI cycles, the couples will then proceed to IVF.
  Interventions: Procedure: intrauterine insemination; Procedure: in vitro fertilization
- II. (Active Comparator): Those randomized to have gonadotropins/IUI treatments first will initiate therapy with two cycles of the fertility injections called FSH or gonadotropins combined with (IUI) intrauterine insemination. If not pregnant after 2 IUI cycles, the couples will then proceed to IVF.
  Interventions: Procedure: intrauterine insemination; Procedure: in vitro fertilization
- III. (Active Comparator): Those couples randomized to (IVF) in vitro fertilization will bypass IUI treatments and start IVF therapy immediately.
  Interventions: Procedure: in vitro fertilization

INTERVENTIONS:
Procedure: intrauterine insemination — An assisted reproduction technique which deposits washed sperm directly into the uterus, bypassing the cervix, and allowing the sperm to enter the fallopian tubes where fertilization normally occurs.
  Other Names: IUI
  Arms: I.; II.
Procedure: in vitro fertilization — This procedure involves stimulating the ovaries, retrieving released eggs, fertilizing the eggs, growing the embryos in a laboratory, and then implanting the embryos in the woman's uterus to develop naturally.
  Other Names: assisted reproductive technologies

SUMMARY:
This study will determine the most effective treatment strategy for infertile couples who present when the female partner is 38 years to the 43rd birthday and the couples are determined to have a reasonable chance for success.

DETAILED DESCRIPTION:
We hypothesize that infertile couples with the female partner 38-43 years of age and demonstrating an adequate ovarian reserve will have higher pregnancy rates at no more cost through immediate IVF than they would through infertility treatment in which IVF is preceded by either two cycles of clomiphene with IUI or two cycles of FSH with IUI.

This hypothesis is being tested by conducting a randomized clinical trial of couples in which the female partner between her 38th and 43rd birthday and determined to have normal ovarian reserve by CCT, and who would otherwise be candidates for ovulation induction/IUI as their initial treatment. The trial will evaluate the efficacy, cost and cost-effectiveness of three alternative infertility treatment strategies: (1) two cycles of clomiphene/IUI followed by IVF, (2) two cycles of FSH/IUI followed by IVF, and (3) immediate IVF; the IVF treatment will include a maximum of four fresh cycles of IVF and two thaw cycles. The trial has the following specific aims:

Aim 1: To compare the proportion of women with a clinically recognized intrauterine pregnancy after two cycles of treatment with clomiphene/IUI, FSH/IUI, or IVF.

Aim 2: To evaluate the overall effectiveness of the three treatment strategies, and their associated complications.

Aim 3: To evaluate the costs and cost effectiveness of the three treatment strategies, including direct and indirect medical costs.

The study participants will be involved in the study for varying amounts of time. The duration of the study will be determined by the treatment cycle in which the participant becomes pregnant. It could be as short as several months' treatment plus the duration of the pregnancy or it could be as long as several years if the participant does not get pregnant or takes breaks during treatment.

This is a collaborative study between Dartmouth College, Boston IVF, Brigham and Women's Hospital, Blue Cross Blue Shield of Massachusetts, Harvard Pilgrim Health Care, and Tufts Health Plan.

Total expected enrollment: 450 Couples

ELIGIBILITY:
Inclusion criteria:

* Female partner age from 38th to the 43rd birthday at the time of recruitment and six months of infertility.
* Male partner has a normal semen analysis showing at least 15 million total motile sperm/ejaculate and at least 1% normal forms by strict criteria, or at least 5 million total motile sperm in an IUI prep.
* Patients must have at least one ovary and at least one ipsilateral patent fallopian tube confirmed by HSG or laparoscopy. Pelvic pathology may be present but must be amenable to operative laparoscopy with the pelvis restored to a functional state, including surgically corrected stages I and II endometriosis. Patients with stage III endometriosis qualify only if the disease is limited to an isolated endometrioma in one or both ovaries and once removed the pelvis is restored to a functional state. For patients with a single patent fallopian tube, the open tube cannot have had a previous ectopic (tubal) pregnancy, and the closed tube cannot be a hydrosalpinx (a tube that is blocked at the end and filled with fluid), unless a cauterization has been performed at the junction of the uterus and fallopian tube. Alternatively, that tube could be removed.
* 4. Normal uterine cavity demonstrated by HSG, sonohysterogram (SHG), or hysteroscopy; pathology of the uterine cavity amenable to operative hysteroscopy (cavity restored to normal and demonstrated by postoperative study).
* Regular menstrual cycles ranging from 21 - 45 days (patients with occasional cycles, i.e. 1 -2 /year, outside this range will be acceptable).
* Acceptable ovarian reserve demonstrated in all patients by a clomiphene challenge test, i.e., cycle day 3 FSH/E2 values of <15 mIU/mL and <100 pg/mL, respectively, and cycle day 10 FSH < 15 mIU/ml. (Note: normal ovarian reserve is represented by FSH values less than 10-12 mIU/mL; our acceptable values represent the transition zone.) Normal TSH and prolactin levels.
* Informed consent from both partners.
* Female body mass index ≤ 38.

Exclusion Criteria:

* Previous tubal or uterine cavity reconstructive surgery in which the pelvis or uterine cavity was not restored to functional.
* Unilateral or bilateral hydrosalpinx (a tube that is blocked at the end and filled with fluid) that has not had a cauterization performed at the junction of the uterus and fallopian tubes, or previous removal of a fallopian tube or an ovary.
* A laparoscopy that demonstrated pelvic adhesions or stage I or II endometriosis for which the pelvis could not be restored to normal by surgery, or endometriosis that was not ablated or excised. All patients with stage IV endometriosis, and those with stage III unless the disease is limited to an isolated endometrioma in one or both ovaries and once removed the pelvis is restored to a functional state.
* One or more prior ectopic pregnancies in which both affected tubes were rendered nonfunctional. One ectopic pregnancy if it existed in the single remaining tube. Two or more ectopic pregnancies even if both tubes are patent.
* Severe male factor (i.e. semen analysis not meeting criteria listed above). Couples using donor semen will be excluded
* Previous treatment with IUI or IVF or for normal ovulatory patients with gonadotropins.
* Inadequate ovarian reserve demonstrating FSH 15 mIU/mL or higher on cycle days 3 or 10 or estradiol 100 pg/mL or higher on cycle day 3.
* Anovulatory patients or those whose cycles are routinely < 21 days or > 45 days in length.
* Patients requiring gamete intrafallopian tube transfer (GIFT), zygote intrafallopian tube transfer (ZIFT), or tubal embryo transfer (TET).
* BMI greater than 38.

Ages: 38 Years to 43 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 450 (Estimated)
Dates: Start 2003-07; Primary Completion 2012-04 (Actual); Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
Associated complications of treatment will be described. | at end of study

SECONDARY OUTCOMES:
Demographics and baseline variables will be collected, including: medical and reproductive, history, age, education, income, race, nutritional history, smoking history, and clinical variables related to infertility diagnosis and treatment. | at end of study

CONTACTS AND LOCATIONS:
Overall Officials: Richard H. Reindollar, M.D., Principal Investigator — Chair, Department of Obstetrics and Gynecology, Dartmouth-Hitchcock Medical Center, Dartmouth Medical School, Lebanon, New Hampshire
Locations (4):
- United States (4):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Boston IVF, Brookline, Massachusetts
  - Boston IVF, Quincy, Massachusetts
  - Boston IVF, Waltham, Massachusetts

REFERENCES:
- [Background] Klipstein S, Regan M, Ryley DA, Goldman MB, Alper MM, Reindollar RH. One last chance for pregnancy: a review of 2,705 in vitro fertilization cycles initiated in women age 40 years and above. Fertil Steril. 2005 Aug;84(2):435-45. doi: 10.1016/j.fertnstert.2005.02.020. PMID 16084887
- [Derived] Nassar KW, Hintzsche JD, Bagby SM, Espinoza V, Langouet-Astrie C, Amato CM, Chimed TS, Fujita M, Robinson W, Tan AC, Schweppe RE. Targeting CDK4/6 Represents a Therapeutic Vulnerability in Acquired BRAF/MEK Inhibitor-Resistant Melanoma. Mol Cancer Ther. 2021 Oct;20(10):2049-2060. doi: 10.1158/1535-7163.MCT-20-1126. Epub 2021 Aug 10. PMID 34376578
- [Derived] Goldman MB, Thornton KL, Ryley D, Alper MM, Fung JL, Hornstein MD, Reindollar RH. A randomized clinical trial to determine optimal infertility treatment in older couples: the Forty and Over Treatment Trial (FORT-T). Fertil Steril. 2014 Jun;101(6):1574-81.e1-2. doi: 10.1016/j.fertnstert.2014.03.012. Epub 2014 Apr 30. PMID 24796764